CLINICAL TRIAL: NCT06838598
Title: Structural and Microbiological Characterization of Arterial Catheter Biofilm in ICU's Patients Using Optical Coherence Tomography
Acronym: OCT-BIO-KTA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier William Morey - Chalon sur Saône (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); Centre Hospitalier Macon (Other)
Responsible Party: Sponsor
Other Study IDs: OCT-BIO-KTA
Record Dates: First submitted 2024-08-21; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Biofilms; Arterial Catheterization, Peripheral; Bacteremia; Tomography, Optical Coherence
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OCT-BIO-KTA cohort: Critically ill patient > 18 years of age with artherial catheter for >2 calendar days in ICU
  Interventions: Other: OCT-BIO-KTA cohort

INTERVENTIONS:
Other: OCT-BIO-KTA cohort — Dynamic full-field optical coherence tomography (D-FF-OCT) analysis of arterial catheter sections before microbiological analysis of catheter biofilm

SUMMARY:
29.3% of bacteremias in intensive care units (ICU) are linked to vascular devices, including 7.7% to arterial catheters, with an influence on both morbility and mortality.

It is now accepted that biofilm as a role on bacterial development on inner surface of vascular devices but there is yet a lack of clinical relevant data documenting a causal relation between biofilm formation and bacteremias.

The investigators assume that a better structural and microbiological characterization of arterial catheter biofilm in ICU patients could help preventing bacteremias or have a more specific treatment when it appears.

ELIGIBILITY:
Inclusion Criteria:

* Patient or relative informed of the study and having declared their non-objection
* Patient over 18 years old
* Patient hospitalized in ICU with an arterial catheter

Exclusion Criteria:

* Patient unable to express consent
* Patient whose collection of the arterial catheter is impossible or for whom storage at 4°C is impossible
* Patient with arterial catheter removed outside the usual procedure of the ICU
* Patient admitted in ICU with an arterial catheter already in place

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years of age with artherial catheter more than 2 calendar days
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Biofilm structure type (ribbon-shaped or mushroom-shaped), measured with D-FF-OCT | Outcome measure is assessed 2 days following catheter removal
  Provide a better understanding of the relation between structural and microbiological characterization of artherial catheter biofilm in ICU patients using D-FF-OCT

SECONDARY OUTCOMES:
Bacterial or fungal indentification | Outcome measure is assessed 2 days following catheter removal
  Identification and enumeration of species - whether bacterial or fungal - by mass spectrometry from culture in agar medium of biofilm samples
Biofilm thickness, measured with D-FF-OCT | Outcome measure is assessed 2 days following catheter removal
  Provide a better understanding of the relation between thickness and microbiological characterization of artherial catheter biofilm in ICU patients using D-FF-OCT
Biofilm dynamic signal distribution, measured with D-FF-OCT | Outcome measure is assessed 2 days following catheter removal
  Provide a better understanding of the relation between dynamic signal distribution and microbiological characterization of artherial catheter biofilm in ICU patients using D-FF-OCT

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Dijon Bourgogne, Dijon, Bourgogne-Franche-Comté
  - CH Macon, Mâcon, Bourgogne-Franche-Comté